CLINICAL TRIAL: NCT06390202
Title: Investigation of the Relationship Between Uterine Artery Doppler Diastolic Notching and Serum Apelin-13 and Apelin-36 Concentrations Between the 11th and 14th Weeks of Pregnancy
Brief Title: Uterine Artery Diastolic Notching & Apelin-13 and 36
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ibrahim kale, associate professor, Umraniye Education and Research Hospital
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/31
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Diagnosis
Keywords: uterine artery; apelin-13; apelin-36; Doppler
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uterine artery notch negative group: Pregnant women who did not have diastolic notching in uterine artery Doppler between the 11th and 14th weeks of pregnancy constituted the uterine artery notch negative group.
  Interventions: Other: no intervention
- Uterine artery notch positive group: Pregnant women with unilateral or bilateral diastolic notching detected in uterine artery Doppler between the 11th and 14th weeks of pregnancy formed the uterine artery notch positive group.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there is no intervention in this study

SUMMARY:
This study was conducted to investigate the relationship between diastolic notching on uterine artery Doppler and serum apelin-13 and 36 concentrations between 11 and 14 weeks of gestation.

DETAILED DESCRIPTION:
Apelin-13 and apelin-36, which provide vasodilatation through a nitric oxide-dependent mechanism, also play a role in trophoblasts' survival, proliferation, and migration.

Based on this, we aimed to investigate serum apelin-13 and apelin-36 concentrations in pregnant women with and without diastolic notch on uterine artery Doppler between the 11th and 14th weeks of pregnancy.

We hypothesized that apelin-13 and apelin-36 might be associated with the formation of diastolic notch in uterine artery Doppler and serum apelin-13 and apelin-36 concentrations would be lower in the group with a notch in the uterine artery Doppler than in the group without a notch.

ELIGIBILITY:
Inclusion Criteria:

1. Nonsmokers,
2. Singleton pregnancies between 11 and 14 weeks of gestation
3. Pregnant women who did not conceive with assisted reproductive methods

Exclusion Criteria:

1. Smokers
2. Pregnant women who conceived with assisted reproductive techniques
3. Pregnant women with multiple pregnancies
4. Pregnant women who started with multiples and continued with singletons
5. Pregnant women with any pregestational disease, thrombophilia
6. Pregnant women with any congenital uterine anomaly
7. Pregnant women with a history of recurrent pregnancy loss
8. Pregnant women using aspirin or heparin

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 44 singleton pregnant women with unilateral or bilateral diastolic notching detected in uterine artery Doppler between the 11th and 14th weeks of pregnancy formed the study group (uterine artery notch positive group). 44 singleton pregnant women who did not have diastolic notching in uterine artery Doppler between the 11th and 14th weeks of pregnancy constituted the control group (uterine artery notch negative group).
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Relationship between diastolic notching on uterine artery Doppler and serum apelin-13 and apelin-36 concentrations. | through study completion, an average of 1 year
  Relationship between diastolic notching on uterine artery Doppler and serum apelin-13 and apelin-36 concentrations.
Relationship between high pulsatility index on uterine artery Doppler and serum apelin-13 and apelin-36 concentrations. | through study completion, an average of 1 year
  Relationship between high pulsatility index on uterine artery Doppler and serum apelin-13 and apelin-36 concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Kale, Associate professor, Study Director — Umraniye Education and Research Hospital
Locations (1):
- Ümraniye Training and Research Hospital, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No